CLINICAL TRIAL: NCT02403440
Title: A Safety, Pharmacokinetics and Pharmacodynamics Study of Hetrombopag Olamine in Chronic Idiopathic Thrombocytopenic Purpura
Brief Title: A Study of Hetrombopag Olamine in Chronic Idiopathic Thrombocytopenic Purpura (ITP) Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPOPId
Record Dates: First submitted 2015-03-20; First posted 2015-03-31 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Purpura, Thrombocytopenic, Idiopathic
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hetrombopag Olamine (Experimental): Hetrombopag Olamine 2.5mg, 5mg and 7.5mg
  Interventions: Drug: Hetrombopag Olamine

INTERVENTIONS:
Drug: Hetrombopag Olamine — Hetrombopag Olamine 2.5mg, 5mg and 7.5mg

SUMMARY:
The purpose of this study is to obtain information on efficacy, safety and Pharmacokinetics (PK)/Pharmacodynamics (PD) of Hetrombopag over 14 days in Chinese patients with chronic ITP.

ELIGIBILITY:
Inclusion Criteria:

1. Chronical ITP patients.
2. The subjects were diagnosed as ITP with bone marrow aspiration within 3 months before enrollment or in the screening period. And secondary immune thrombocytopenia (e.g., myelodysplastic syndrome, systemic lupus erythematosus, aplastic anemia) was excluded.
3. Patients had a mean platelet count of less than 30,000/µL in the screening period.
4. Patients receiving chronic maintenance steroid therapy must have received a stable dose for at least 1 month.
5. Patients receiving danazol, mycophenolate mofetil or cyclosporine A must have received a stable dose for at least 12 weeks.
6. Normal PT/INR and APTT.

Exclusion Criteria:

1. Any prior history of arterial or venous thrombosis (stroke, transient ischemic attack, myocardial infarction, deep vein thrombosis or pulmonary embolism), AND ≥ two of the following risk factors: hormone replacement therapy, systemic contraception (containing estrogen), smoking, diabetes, hypercholesterolemia, medication for hypertension, cancer, hereditary thrombophilic disorders (e.g., Factor V Leiden, ATIII deficiency, etc), or any other family history of arterial or venous thrombosis.
2. Pre-existing cardiovascular disease (congestive heart failure, New York Heart Association [NYHA] Grade III/IV), or arrhythmia known to increase the risk of thromboembolic events (e.g. atrial fibrillation).
3. Malignant disease
4. Cancer treatment with cytotoxic chemotherapy and/or radiotherapy.
5. Patients with one of the following conditions should be excluded:

   * Treatment with immunoglobulins within 1 week preceding the first dose of study medication.
   * Treatment with splenectomy or rituximab within 12 weeks preceding the first dose of study medication.
   * Treatment with eltrombopag or Nplate within 4 weeks preceding the first dose of study medication.
   * Treatment with cyclophosphamide or vinca alkaloids within 4 weeks preceding the first dose of study medication.
6. ALT>2×ULN，AST>2×ULN，Total Bilirubin>1.5×ULN，serum creatinine >1.2×ULN，Total albumin <0.9×LLN

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
The number of volunteers with adverse events as a measure of safety and tolerability | up to Day 28

SECONDARY OUTCOMES:
Plasma pharmacokinetic (PK) parameters of Hetrombopag after multiple dose from day 1 to day 14, composite including AUC, Cmax, Tmax, and t1/2 | day 1 and day 14
The proportion of patients with platelet counts ≥50,000/µL after treatment | up to Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- West Hospital, Sichuan University, Chengdu, China

REFERENCES:
- [Derived] Wang Z, Chen L, Zhang F, Lu H, Chen X, Wen A, Luo J, Hu Y, Wang Y, Niu T, Zheng L. First-in-patient study of hetrombopag in patients with chronic idiopathic thrombocytopenic purpura. J Thromb Haemost. 2020 Nov;18(11):3053-3060. doi: 10.1111/jth.15078. Epub 2020 Oct 1. PMID 32865293